CLINICAL TRIAL: NCT06809660
Title: Effects of Endocrine Disruptors on the Gut Microbiota and Assessment of Their Impact on Colorectal Cancer Development
Brief Title: Effects of Endocrine Disruptors on the Gut Microbiota and Assessment of Their Impact on Colorectal Cancer Development (PERMICA)
Acronym: PERMICA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Collaborators: University of Poitiers - Laboratoire Ecologie et Biologie des Interactions (EBI) - UMR CNRS 7267 (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-A02197-40
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Cancer (CRC); Endocrine Disruptors; Microbiota; Dysbiosis
MeSH Terms: conditions — Colorectal Neoplasms; Dysbiosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient with colorectal cancer (Other)
  Interventions: Other: Collection of biological samples and clinical data
- Patient without suspected colorectal cancer (Other)
  Interventions: Other: Collection of biological samples and clinical data

INTERVENTIONS:
Other: Collection of biological samples and clinical data — * Collection of a hair sample
  * Collection of urine
  * Collection of stool samples
  * Collection of clinical, paraclinical data, and exposure questionnaire

SUMMARY:
Colorectal cancer is the third most common cancer worldwide, yet it was the second leading cause of cancer-related deaths in 2020. The average French population faces a colorectal cancer risk partly linked to lifestyle factors. The majority of colorectal cancer cases (approximately 85%) are not caused by hereditary mutations. Environmental factors, such as lifestyle or diet (notably through endocrine disruptors), can affect the gut microbiota (a collection of microorganisms - bacteria, viruses, parasites, and fungi - residing in the intestinal environment) and lead to disturbances in its composition, referred to as dysbiosis. While the mechanisms underlying dysbiosis associated with colorectal cancer remain poorly understood, the involvement of certain ingested substances, known as xenobiotics, is increasingly suspected, including endocrine disruptors. Among the most common endocrine disruptors found in water and food are parabens and phthalates, which will be examined in detail in this study. These substances may be directly involved in the development of colorectal cancer and in response to its treatment.

The main objective of this studie is to characterize the relationship between colorectal cancer diagnosis, activity/composition of the gut microbiota, and patients' exposure to selected endocrine disruptors, particularly parabens and phthalates.

DETAILED DESCRIPTION:
Methodology:

Pilot, single-center regional study, with a descriptive and comparative design (patients with colorectal cancer / patients without suspected colorectal cancer = controls).

In each group, a stool, hair and urine sample will be collected and an endocrine disruptor exposure questionnaire completed.

Sample Size and Duration:

A total of 200 patients will be included, divided into two groups of 100 patients (100 patients with colorectal cancer and 100 patients without suspected colorectal cancer). The inclusion period will last 48 months, with each participant enrolled for a maximum of one month. Routine care data will be collected over 5 years. The total duration of the clinical investigation will be approximately 9 years.

Expected Outcomes:

The investigators aim at determining whether the most common endocrine disruptors in the French population are involved in colorectal carcinogenesis and if these substances are correlated with dysbiotic colorectal microbiota.

The findings from this study should help identify the endocrine disruptors most frequently associated with colorectal cancer and thereby enhance vigilance regarding these substances.

Benefits for Patients:

There are no individual but collective benefits, as the results will colorectal cancer related knowledge and its relationship with lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled endoscopy during the inclusion visit or within 18 months following this consultation.
* Signed consent from the patient after clear and fair information about the study is provided.
* Patient is free of guardianship, curatorship, or dependency.
* Patient is covered by a social security system or through a third party.

Exclusion Criteria:

* Patients receiving treatment for chronic inflammatory bowel disease;
* Patients with hereditary colorectal cancer;
* Use of antibiotics, probiotics, or prebiotics within four weeks prior to stool sample collection;
* Patients who have undergone neoadjuvant chemotherapy or radiotherapy;
* Patients who have had previous surgical resection;
* Patients under enhanced protection: minors, individuals deprived of liberty by judicial or administrative decision, individuals residing in healthcare or social institutions, and adults under legal protection;
* Pregnant and/or breastfeeding women.

Exclusion Criteria During Study Participation:

* Patients presenting any of the following during their participation in the study will be excluded:
* Use of antibiotics, probiotics, or prebiotics before stool collection (between inclusion and stool collection, which may occur within the month);
* Endoscopy not performed within 18 months following inclusion;
* Failure to send/receive stool samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2031-01-21 (Estimated); Study Completion 2034-01-21 (Estimated)

PRIMARY OUTCOMES:
Association between faecal microbiota disruption and exposure to endocrine disruptors | 1 month/patient (maximum time between enrolment visit and stool collection)
  Association between disruptions in the composition and/or activity of the faecal microbiota (sequencing and metabolome analysis) and exposure to endocrine disruptors (measured in urine and stool samples) in patients with colorectal cancer and in controls

SECONDARY OUTCOMES:
Describe the accumulated exposome | 1 day/patient
  LC/MS on hair samples
Describe gut microbiota composition | 1 month/patient (maximum time between enrolment visit and stool collection)
  From stool samples
Detect differences in pro-carcinogenic bacteria | 1 month/patient (maximum time between enrolment visit and stool collection)
  In stool samples
Correlation metabolome / gut microbiota in patients with colorectal cancer | 1 month/patient (maximum time between enrolment visit and stool collection)
  Analysis of the correlation between the metabolome and gut microbiota in colorectal cancer patients

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No